CLINICAL TRIAL: NCT01622608
Title: Adolescent Vaccination Kiosk Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Society for Adolescent Health & Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-0179
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Adolescent Vaccination Status
Keywords: Adolescent vaccination; Immunization rates; Informational kiosk; Tailored health messaging; Barriers to vaccination; Attitudes; Intentions
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kiosk Users (Experimental)
  Interventions: Behavioral: Vaccine Information Kiosk
- Non-Kiosk Users (No Intervention)

INTERVENTIONS:
Behavioral: Vaccine Information Kiosk — The study kiosk will remain in the waiting room of participating practices for the duration of the study. Interested parents will self-direct to the kiosk in the clinic waiting room either before or after their child's appointment. Following consent, parents will complete a survey that assesses socio-demographics, baseline vaccination intention, and vaccine-specific beliefs, attitudes and experiences. The kiosk will generate tailored educational messages about adolescent vaccines. Parents can utilize the kiosk as many times as they wish during the intervention period.
  Arms: Kiosk Users

SUMMARY:
The purpose of this study is to determine whether implementation of a web-based educational intervention using a "vaccine information kiosk" placed in primary care practice waiting rooms can reach a large number of parents and have a measurable impact on adolescent vaccination rates, specifically for Tdap, HPV, meningococcal, and influenza vaccines.

DETAILED DESCRIPTION:
Adolescents are a reservoir population for a variety of vaccine preventable diseases (VPDs). Despite this, adolescent vaccination rates lag substantially behind national goals of 80% coverage for adolescent vaccines set forth by Healthy People 2020. This has been particularly the case for the vaccines most recently recommended for adolescents, such as the human papillomavirus (HPV) and seasonal influenza (flu) vaccines; national coverage levels in 2010 for HPV were 32% (for series completion among females only) and 35% for flu vaccine. Uptake levels for the two other adolescent-targeted vaccines, tetanus-diphtheria-acellular pertussis (Tdap) and meningococcal conjugate (MCV4) vaccines are currently at 69% and 63%, respectively.

A major barrier to increased adolescent vaccination levels is the lack of parental and provider recognition that an adolescent is due for vaccine doses. For providers, there are the dual challenges of getting adolescents to come in for annual preventive care visits and also minimizing "missed opportunities" for vaccination (i.e. clinical interactions with a patient where a needed vaccine could have been provided but was not). Reminder/recall systems are one mechanism to help address both of these challenges for providers while also informing parents about the need for adolescent vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Parents of adolescents (11-17 years) attending one of 3 participating pediatric practices.
* able to read and converse in English.

Exclusion Criteria:

* Parent age < 18 years,
* prisoners,
* decisionally challenged participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Utilization of vaccine information kiosks by parents/patients. | 12 months
  Descriptive statistics on kiosk utilization patterns overall, and disaggregated by various demographic, attitudinal and vaccination status categories will be derived. This will be assessed in intervention settings using data entered by parents, as well as paradata such as the order of web pages viewed, and time spent per page.
Usefulness of vaccine information kiosks | 12 months (provider survey) & 3 months (parent survey)
  Parent satisfaction with the material presented in the kiosk, as well as changes between parents' baseline survey (done at the kiosk) and follow-up email survey in: 1) parent attitudes about vaccination and 2) parent vaccine-specific vaccination intention will be assessed. Provider views on having the kiosks in the waiting room of their clinic will also be assessed.
Proportion of adolescents who had a change in their vaccination status in kiosk users compared to non-users. | 12 months
  Vaccination status will be determined primarily by medical record review, and augmented by parent report. The proportion of adolescents who had a change in their vaccination status (Tdap, MCV, HPV, Flu) before versus after their clinic visit (for non-users of the kiosk), or before versus after the date their parent first accessed the intervention (for users of the kiosk) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Dempsey, MD, PhD, MPH, Principal Investigator — University of colorado, Children's Hospital Colorado; Sean O'Leary, MD, MPH, Principal Investigator — University of Colorado Denver, Children's Hospital Colorado; Lawrence An, MD, Principal Investigator — University of Michigan, Masonic Cancer Center
Locations (3):
- United States (3):
  - Pediatrics 5280, Centennial, Colorado
  - Mountainland Pediatrics, Thornton, Colorado
  - Pediatrics West, Wheat Ridge, Colorado